CLINICAL TRIAL: NCT01605227
Title: A Phase 3, Randomized, Double-blind, Controlled Study of Cabozantinib (XL184) Versus Prednisone in Metastatic Castration-resistant Prostate Cancer Patients Who Have Received Prior Docetaxel and Prior Abiraterone or MDV3100
Brief Title: Study of Cabozantinib (XL184) Versus Prednisone in Men With Metastatic Castration-resistant Prostate Cancer Previously Treated With Docetaxel and Abiraterone or MDV3100
Acronym: COMET-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XL184-307; 2012-001834-33 (EudraCT Number)
Record Dates: First submitted 2012-05-22; First posted 2012-05-24 (Estimated); Results first posted 2018-03-14 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2018-02

CONDITIONS: Prostate Cancer; Castration Resistant Prostate Cancer; Pain; Prostatic Neoplasms
Keywords: prostate cancer; castration resistant prostate cancer; bone pain; CRPC
MeSH Terms: conditions — Prostatic Neoplasms; Pain | interventions — cabozantinib; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cabozantinib (Experimental): Subjects randomized to the cabozantinib arm will also receive placebo-matched prednisone capsules.
  Interventions: Drug: cabozantinib
- prednisone (Active Comparator): Subjects randomized to the prednisone arm will also receive placebo-matched cabozantinib.
  Interventions: Drug: prednisone

INTERVENTIONS:
Drug: cabozantinib — Tablets taken orally once-daily
  Other Names: XL184
  Arms: cabozantinib
Drug: prednisone — Taken twice a day orally. Commercially-obtained prednisone tablets will be over-encapsulated in order to blind identity.
  Arms: prednisone

SUMMARY:
This study will evaluate the effect of cabozantinib compared to prednisone on overall survival in men with previously treated metastatic castration-resistant prostate cancer with bone-dominant disease who have experienced disease progression on docetaxel-containing chemotherapy and abiraterone or MDV3100.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of castration resistant prostate cancer (serum testosterone less than 50 ng/dL).
* Evidence of bone metastasis related to prostate cancer on bone scans.
* Received prior docetaxel (minimum cumulative dose of 225 mg/m2) and either abiraterone or MDV3100 treatment and has evidence of prostate cancer progression on each agent independently.
* Maintenance of LHRH agonist or antagonist unless treated with orchiectomy.
* Recovered from toxicities related to any prior treatments, unless the toxicities are clinically non significant or easily manageable.
* Adequate organ and marrow function.
* Capable of understanding and complying with the protocol requirements and signed the informed consent form.
* Sexually active fertile patients and their partners must agree to use medically accepted methods of contraception (eg, barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for 4 months after the last dose of study treatment.

Exclusion Criteria:

* Prior treatment with cabozantinib.
* Treatment with docetaxel, abiraterone, or MDV3100 in the last 2 weeks; or with any other type of cytotoxic or investigational anticancer agent in the last 2 weeks.
* Radiation within 4 weeks (excluded if to mediastinum) or radionuclide treatment within 6 weeks of randomization.
* Known brain metastases or cranial epidural disease.
* Requires concomitant treatment, in therapeutic doses, with anticoagulants.
* Requires chronic concomitant treatment of strong CYP3A4 inducers (eg, dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbital, and St. John's Wort).
* Uncontrolled, significant intercurrent illness including, but not limited to, cardiovascular disorders, gastrointestinal disorders, active infections, non-healing wounds, recent surgery.
* Clinically significant hematemesis or hemoptysis, or other signs indicative of pulmonary hemorrhage in the last 3 months, or history of other significant bleeding in the past 6 months.
* Cavitating pulmonary lesion(s) or a lesion invading or encasing a major blood vessel.
* QTcF > 500 ms within 7 days of randomization.
* Unable to swallow capsules or tablets.
* Previously-identified allergy or hypersensitivity to components of the study treatment formulations.
* Another diagnosis of malignancy requiring systemic treatment within 2 years of randomization.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1028 (Actual)
Dates: Start 2012-07; Primary Completion 2014-09 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (238):
- United States (76):
  - Birmingham, Alabama
  - Anchorage, Alaska
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Jonesboro, Arkansas
  - Duarte, California
  - Highland, California
  - La Jolla, California
  - Los Angeles, California
  - Montebello, California
  - Orange, California
  - Palo Alto, California
  - Rancho Mirage, California
  - San Marcos, California
  - St. Helena, California
  - Vallejo, California
  - Aurora, Colorado
  - New Haven, Connecticut
  - Southington, Connecticut
  - Miami Beach, Florida
  - Ocala, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Titusville, Florida
  - Wellington, Florida
  - West Palm Beach, Florida
  - Athens, Georgia
  - Atlanta, Georgia
  - Marietta, Georgia
  - Galesburg, Illinois
  - Niles, Illinois
  - Ames, Iowa
  - Sioux City, Iowa
  - Wichita, Kansas
  - Hazard, Kentucky
  - Louisville, Kentucky
  - Brewer, Maine
  - Baltimore, Maryland
  - Bethesda, Maryland
  - Towson, Maryland
  - Boston, Massachusetts
  - Methuen, Massachusetts
  - Detroit, Michigan
  - Wyoming, Michigan
  - Minneapolis, Minnesota
  - Jefferson City, Missouri
  - Springfield, Missouri
  - Lincoln, Nebraska
  - Omaha, Nebraska
  - Hackensack, New Jersey
  - Lawrenceville, New Jersey
  - Albany, New York
  - Garden City, New York
  - New York, New York
  - Pinehurst, North Carolina
  - Bismarck, North Dakota
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Portland, Oregon
  - Bryn Mawr, Pennsylvania
  - Hershey, Pennsylvania
  - Lancaster, Pennsylvania
  - Greenville, South Carolina
  - Chattanooga, Tennessee
  - Amarillo, Texas
  - Bedford, Texas
  - Houston, Texas
  - Laredo, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Burlington, Vermont
  - Fairfax, Virginia
  - Newport News, Virginia
  - Spokane, Washington
  - Green Bay, Wisconsin
- Australia (18):
  - Albury, New South Wales
  - Concord, New South Wales
  - Darlinghurst, New South Wales
  - Kogarah, New South Wales
  - Port Macquarie, New South Wales
  - Randwick, New South Wales
  - Wahroonga, New South Wales
  - Westmead, New South Wales
  - South Brisbane, Queensland
  - Southport, Queensland
  - Woolloongabba, Queensland
  - Adelaide, South Australia
  - Kurralta Park, South Australia
  - Hobart, Tasmania
  - Bentleigh East, Victoria
  - Box Hill, Victoria
  - Wodonga, Victoria
  - Perth, Western Australia
- Austria (4):
  - Linz
  - Salzburg
  - Vienna
  - Wein
- Belgium (8):
  - Aalst
  - Bonheiden
  - Brussels
  - Ghent
  - Hasselt
  - Leuven
  - Liège
  - Roeselare
- Canada (8):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Miramichi, New Brunswick
  - Halifax, Nova Scotia
  - London, Ontario
  - Owen Sound, Ontario
  - Montreal, Quebec
  - Québec
- France (19):
  - Angers
  - Besançon
  - Bordeaux
  - Caen
  - Clermont-Ferrand
  - Dijon
  - La Roche-sur-Yon
  - Le Mans
  - Lille
  - Lyon
  - Marseille
  - Nancy
  - Paris
  - Pierre-Bénite
  - Rennes
  - Saint-Herblain
  - Strasbourg
  - Suresnes
  - Villejuif
- Germany (26):
  - Aachen
  - Berlin
  - Braunschweig
  - Cologne
  - Dresden
  - Düsseldorf
  - Frankfurt am Main
  - Freiburg im Breisgau
  - Fürth
  - Gütersloh
  - Hamburg
  - Hanover
  - Heidelberg
  - Homburg
  - Kassel
  - Kempen
  - Kirchheim
  - Mannheim
  - München
  - Münster
  - Nürtingen
  - Offenburg
  - Traunstein
  - Tübingen
  - Weiden
  - Wuppertal
- Ireland (3):
  - Cork
  - Dublin
  - Galway
- Italy (24):
  - Ancona
  - Arezzo
  - Aviano
  - Brindisi
  - Cremona
  - Genova
  - Livorno
  - Meldola
  - Milan
  - Modena
  - Napoli
  - Novara
  - Orbassano
  - Padua
  - Pavia
  - Pisa
  - Pordenone
  - Ravenna
  - Rimini
  - Roma
  - Rozzano
  - Terni
  - Torino
  - Verona
- Netherlands (8):
  - Amsterdam
  - Groningen
  - Hoofddorp
  - Nieuwegein
  - Nijmegen
  - Rotterdam
  - Tilburg
  - Zwolle
- Ponce, Puerto Rico
- Spain (16):
  - Málaga, Andalusia
  - Seville, Andalusia
  - Palma de Mallorca, Balearic Islands
  - San Cristóbal de La Laguna, Canary Islands
  - Badalona, Catalonia
  - Barcelona, Catalonia
  - L'Hospitalet de Llobregat, Catalonia
  - Manresa, Catalonia
  - A Coruña, Galicia
  - Santiago de Compostela, Galicia
  - Madrid, Madrid, Communidad de
  - Majadahonda, Madrid, Communidad de
  - Pamplona, Navarre
  - Oviedo, Principality of Asturias
  - Elche, Valencia
  - Valencia, Valencia
- Sweden (7):
  - Gotenborg
  - Malmo
  - Örebro
  - Stockholm
  - Umeå
  - Uppsala
  - Vaxjo
- United Kingdom (20):
  - Aberdeen
  - Bath
  - Birmingham
  - Brighton
  - Bristol
  - Cambridge
  - Cardiff
  - Cottingham
  - Edinburgh
  - Inverness
  - Lancaster
  - Leeds
  - London
  - Maidstone
  - Metropolitan Borough of Wirral
  - Northwood
  - Plymouth
  - Sheffield
  - Southampton
  - Sutton

REFERENCES:
- [Derived] Heller G, McCormack R, Kheoh T, Molina A, Smith MR, Dreicer R, Saad F, de Wit R, Aftab DT, Hirmand M, Limon A, Fizazi K, Fleisher M, de Bono JS, Scher HI. Circulating Tumor Cell Number as a Response Measure of Prolonged Survival for Metastatic Castration-Resistant Prostate Cancer: A Comparison With Prostate-Specific Antigen Across Five Randomized Phase III Clinical Trials. J Clin Oncol. 2018 Feb 20;36(6):572-580. doi: 10.1200/JCO.2017.75.2998. Epub 2017 Dec 22. PMID 29272162
- [Derived] Smith M, De Bono J, Sternberg C, Le Moulec S, Oudard S, De Giorgi U, Krainer M, Bergman A, Hoelzer W, De Wit R, Bogemann M, Saad F, Cruciani G, Thiery-Vuillemin A, Feyerabend S, Miller K, Houede N, Hussain S, Lam E, Polikoff J, Stenzl A, Mainwaring P, Ramies D, Hessel C, Weitzman A, Fizazi K. Phase III Study of Cabozantinib in Previously Treated Metastatic Castration-Resistant Prostate Cancer: COMET-1. J Clin Oncol. 2016 Sep 1;34(25):3005-13. doi: 10.1200/JCO.2015.65.5597. Epub 2016 Jul 11. PMID 27400947

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled: 02 July 2012 (first subject randomized), Data cut off date: 07 July 2014
Groups:
- Cabozantinib: Subjects randomized to the cabozantinib arm will also receive placebo-matched prednisone capsules.
  Cabozantinib (XL184) 60 mg tablets orally once daily plus prednisone-matched placebo orally twice daily.
- Prednisone: Subjects randomized to the prednisone arm will also receive placebo-matched cabozantinib.
  Prednisone 5 mg capsules orally twice daily plus cabozantinib-matched placebo orally once daily.
Period: Overall Study
Arm/Group | Cabozantinib | Prednisone
Started (Randomized) | 682 | 346
Completed (Subjects still on study treatment at data cut-off date) | 61 | 17
Not Completed | 621 | 329
Not completed — Did not receive study treatment | 2 | 3
Not completed — Adverse Event | 228 | 42
Not completed — Progressive Disease | 132 | 128
Not completed — Clinical Deterioration | 227 | 133
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Physician Decision | 9 | 7
Not completed — Withdrawal by Subject | 18 | 14
Not completed — Sponsor Decision | 2 | 0
Not completed — Started New Therapy | 1 | 0
Not completed — Subject Decision | 0 | 1
Not completed — Dose Held >6 weeks | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cabozantinib | Prednisone | Total
Number analyzed (Participants) | 682 | 346 | 1028
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 165 | 97 | 262
  >=65 years | 517 | 249 | 766
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 682 | 346 | 1028
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 6 | 20
  White | 520 | 265 | 785
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 146 | 74 | 220
Region of Enrollment [Count of Participants; unit: Participants]
  North America | 119 | 63 | 182
  Europe | 528 | 256 | 784
  Australia | 35 | 27 | 62
Prior cabazitaxel (per CRF) [Count of Participants; unit: Participants]
  Yes | 261 | 132 | 393
  No | 421 | 214 | 635
Brief Pain Inventory (BPI) Item 3 (per CRF) [Count of Participants; unit: Participants] — Pain will be assessed using the BPI Items #3 (worst pain over the last 24 hours by recall).
  Participants
    <4 | 389 | 196 | 585
    ≥4 | 284 | 148 | 432
    Missing | 9 | 2 | 11
ECOG Performance Status (per CRF) [Number; unit: participants]
  0/1 (asymptomatic or symptomatic but ambulatory) | 605 | 303 | 908
  2 (ambulatory but can't carry out work activities) | 76 | 43 | 119
  Missing | 1 | 0 | 1
Opioid narcotic use within 24 hours (per solicited oploid CRF) [Count of Participants; unit: Participants] | 454 | 228 | 682
Concomitant prednisone/prednisolone at randomization [Count of Participants; unit: Participants] | 289 | 142 | 431
Time from diagnosis to study entry [Median (Full Range); unit: years] | 6.68 [0.09 to 26.6] | 6.98 [0.04 to 22.2] | 6.83 [0.04 to 26.6]
Bone scan lesion area [Median (Full Range); unit: mm^2] | 45,635.5 [0 to 388,052] | 41,746.0 [0 to 283,304] | 44,782.0 [0 to 388,052]
Extent of metastasis [Number; unit: participants]
  None | 0 | 0 | 0
  Bone | 681 | 346 | 1027
  Lymph node | 313 | 140 | 453
  Visceral | 133 | 58 | 191
  Liver | 91 | 35 | 126
  Lung | 69 | 29 | 98
  Other soft tissue | 39 | 23 | 62
No. of prior anticancer agents [Number; unit: participants] — Excluding agents to maintain castration status
  participants
    2 | 57 | 31 | 88
    ≥3 | 625 | 315 | 940
Baseline LDH [Median (Full Range); unit: U/L] | 230 [59 to 6004] | 230 [87 to 3062] | 230 [59 to 6004]
Baseline PSA [Median (Full Range); unit: μg/L] | 192 [0.02 to 10030] | 195 [0.54 to 10963] | 192 [0 to 10963]
Baseline serum testosterone (<50 ng/dL) [Count of Participants; unit: Participants] | 677 | 345 | 1022

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: The primary analysis of OS is defined as the time from randomization to death due to any cause. Participants that had not died or were permanently lost to follow-up were censored at the last known date alive. Median OS was calculated using Kaplan-Meier estimates. Analysis for OS was performed after 614 events had occurred.
Time Frame: OS was measured from the time of randomization until 614 events, approximately 24 months after study start
Population: The Intent to Treat (ITT) population was used and included 1028 randomized subjects (682 cabozantinib, 346 prednisone).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabozantinib | Prednisone
Number analyzed (Participants) | 682 | 346
months | 11.0 [10.09 to 11.63] | 9.8 [9.00 to 11.53]
Statistical Analysis 1: Comparison: Cabozantinib vs Prednisone; Test type: Superiority or Other; p = 0.213, Log Rank; The Log-Rank test was stratified by prior cabazitaxel, baseline pain severity and baseline ECOG performance status; Cox Proportional Hazard = 0.90, 95% CI 2-sided [0.76 to 1.06]

2. Secondary Outcome: Bone Scan Response (BSR)
Description: BSR is defined as >=30% reduction in the bone scan lesion area (BSLA) compared with baseline. Confirmation of bone scan was not required for response or progression. Bone scans were evaluated by an independent radiology facility (IRF) for response.
Time Frame: BSR was measured at the end of Week 12 as determined by the IRF
Population: Analysis was conducted on the ITT population (682 cabozantinib, 346 prednisone) for Bone Scan Response (BSR) at Week 12.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cabozantinib | Prednisone
Number analyzed (Participants) | 682 | 346
percentage of participants | 42 [38 to 46] | 3 [1 to 5]
Statistical Analysis 1: Comparison: Cabozantinib vs Prednisone; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; The Cochran-Mantel-Haenszel (CMH) Test was stratified by prior cabazitaxel, baseline pain severity and baseline ECOG performance status

3. Other Pre Specified Outcome: Progression-free Survival (PFS)
Description: The exploratory analysis of PFS is the time from randomization to date of first documented radiographic progression (bone and/or soft tissue) according to the investigator's assessment or death. PFS was defined per mRECIST 1.1 and included evaluation of measurable, nonmeasurable, target and nontarget lesions. A Kaplan-Meier analysis was performed to estimate the median duration.
Time Frame: Duration of PFS was defined as time from the date of randomization to earlier of date of radiographic progression (bone/andor soft tissue) according to the investigator's assessment or death, assessed for up to approximately 24 months
Population: The Intent to Treat (ITT) population was used and include 1028 randomized subjects (682 cabozantinib, 346 prednisone) with a data cut off date of 07 July 2014.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabozantinib | Prednisone
Number analyzed (Participants) | 682 | 346
months | 5.6 [5.49 to 5.62] | 2.8 [2.79 to 2.86]
Statistical Analysis 1: Comparison: Cabozantinib vs Prednisone; Test type: Superiority or Other; p < 0.001, Log Rank; The Log-Rank Test was stratified by prior cabazitaxel, baseline pain severity, and baseline Eastern Cooperative Oncology Group Performance Status; Hazard Ratio (HR) = 0.48, 95% CI 2-sided [0.40 to 0.57]

ADVERSE EVENTS:
Time Frame: Up to 92 weeks
Description: Safety was assessed based on the date of first dose and at minimum every 3 weeks up to Week 12 and every 6 weeks thereafter. The safety data includes subjects who were randomized and treated. Of 1028 patients, 682 were randomized to receive cabozantinib and 346 prednisone. The Safety population comprised of 1023 patients (681 cabozantinib, 342 prednisone).
Arm/Group | Cabozantinib | Prednisone
Serious Adverse Events (participants affected / at risk) | 420/681 | 181/342
Other Adverse Events (participants affected / at risk) | 675/681 | 332/342
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cabozantinib (N=681) | Prednisone (N=342)
Anaemia (Blood and lymphatic system disorders) | 32 | 16
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Pancytopenia (Blood and lymphatic system disorders) | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 4
Acute coronary syndrome (Cardiac disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 5 | 0
Angina pectoris (Cardiac disorders) | 2 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 5 | 2
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 4 | 1
Cardiac failure congestive (Cardiac disorders) | 2 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 1
Cystic lymphangioma (Congenital, familial and genetic disorders) | 1 | 0
Metabolic myopathy (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Cushing's syndrome (Endocrine disorders) | 1 | 0
Hypoaldosteronism (Endocrine disorders) | 1 | 0
Diplopia (Eye disorders) | 1 | 1
Visual acuity reduced (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 8 | 3
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 2 | 0
Anal inflammation (Gastrointestinal disorders) | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 12 | 6
Diarrhoea (Gastrointestinal disorders) | 10 | 2
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enterovesical fistula (Gastrointestinal disorders) | 1 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 2 | 0
Gastric antral vascular estasia (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 2 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 | 0
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 3 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 23 | 6
Obstruction gastric (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstrucion (Gastrointestinal disorders) | 1 | 0
Small intestinal perforation (Gastrointestinal disorders) | 2 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 28 | 6
Asthenia (General disorders) | 18 | 3
Chest pain (General disorders) | 2 | 0
Death (General disorders) | 4 | 1
Device dislocation (General disorders) | 1 | 0
Device occlusion (General disorders) | 1 | 0
Drug withdrawal syndrome (General disorders) | 1 | 0
Euthanasia (General disorders) | 3 | 0
Fatigue (General disorders) | 20 | 3
General physical health deterioration (General disorders) | 52 | 22
Influenza like illness (General disorders) | 1 | 0
Local swelling (General disorders) | 2 | 1
Malaise (General disorders) | 5 | 0
Mucosal inflammation (General disorders) | 8 | 0
Multi-organ failure (General disorders) | 2 | 2
Non-cardiac chest pain (General disorders) | 2 | 1
Oedema peripheral (General disorders) | 3 | 1
Pain (General disorders) | 10 | 7
Performance status decreased (General disorders) | 1 | 0
Pyrexia (General disorders) | 15 | 6
Sudden death (General disorders) | 1 | 1
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Hepatic failure (Hepatobiliary disorders) | 3 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hydrocholecystis (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0
Abdominal sepsis (Infections and infestations) | 1 | 0
Abscess (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 4 | 0
Appendicitis (Infections and infestations) | 1 | 0
Arthritis infective (Infections and infestations) | 1 | 0
Aspergillus infection (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Colonic abscess (Infections and infestations) | 3 | 0
Cystitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 2
Device related sepsis (Infections and infestations) | 2 | 1
Endocarditis (Infections and infestations) | 1 | 0
Endocarditis staphylococcal (Infections and infestations) | 1 | 0
Enterobacter infection (Infections and infestations) | 1 | 0
Enterobactar sepsis (Infections and infestations) | 0 | 1
Enterococcal sepsis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 3 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 1
Lung infection (Infections and infestations) | 5 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Osteomyelilitis (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0
Periorbital cellulitis (Infections and infestations) | 1 | 0
Pharyngeal abscess (Infections and infestations) | 1 | 0
Pilonidal cyst (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 17 | 12
Pneumonia klebsiella (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 2 | 0
Pulpitis dental (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 3 | 0
Sepsis (Infections and infestations) | 11 | 5
Septic shock (Infections and infestations) | 3 | 2
Sinusitis (Infections and infestations) | 1 | 0
Spinal cord infection (Infections and infestations) | 1 | 5
Staphylococcal infection (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 2 | 1
Streptococcal bacteraemia (Infections and infestations) | 1 | 1
Streptococcal infection (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 13 | 6
Urinary tract infection enterococcal (Infections and infestations) | 0 | 1
Urinary tract infection staphylococcal (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 7 | 1
Viral infection (Infections and infestations) | 0 | 1
Viral pharyngitis (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Chest injury (Injury, poisoning and procedural complications) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Keratorhexis (Injury, poisoning and procedural complications) | 1 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Urostomy complication (Injury, poisoning and procedural complications) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Blood creatine increased (Investigations) | 2 | 0
Clostridium test positive (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 2
Platelet count decreased (Investigations) | 1 | 0
Red blood cell count decreased (Investigations) | 0 | 1
Troponin T increased (Investigations) | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 15 | 2
Dehydration (Metabolism and nutrition disorders) | 20 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 2 | 1
Hyperglyceaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 7 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 15 | 11
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 4 | 4
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Hormone-refractory prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 3
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 19 | 12
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nodular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 52 | 27
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cauda equina syndrome (Nervous system disorders) | 1 | 1
Cerebellar infarction (Nervous system disorders) | 1 | 0
Cerebral haematoma (Nervous system disorders) | 2 | 0
Cerebral haemorrhage (Nervous system disorders) | 3 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 2 | 1
Cerebrovascular accident (Nervous system disorders) | 4 | 3
Cognitive disorder (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 2 | 0
Dyskinesia (Nervous system disorders) | 1 | 0
Facial paresis (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 3
Hemiparesis (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 4
Ischaemic stroke (Nervous system disorders) | 1 | 1
Lethargy (Nervous system disorders) | 2 | 0
Leukoencephalopathy (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 3 | 1
Memory impairment (Nervous system disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Nerve root compression (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Paraparesis (Nervous system disorders) | 0 | 2
Paralpegia (Nervous system disorders) | 0 | 2
Parkinson's disease (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 1
Quadriparesis (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Sensorimotor disorder (Nervous system disorders) | 0 | 1
Sensory loss (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 14 | 8
Spinal cord paralysis (Nervous system disorders) | 0 | 1
Stupor (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 5 | 2
Agitation (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1
Confusional state (Psychiatric disorders) | 7 | 0
Delirium (Psychiatric disorders) | 2 | 1
Depression (Psychiatric disorders) | 0 | 1
Bladder dysfunction (Renal and urinary disorders) | 0 | 1
Bladder outlet obstruction (Renal and urinary disorders) | 0 | 1
Calculus bladder (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 5 | 3
Hydronephrosis (Renal and urinary disorders) | 5 | 4
Hydroureter (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Prerenal failure (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 2 | 3
Renal failure acute (Renal and urinary disorders) | 12 | 4
Renal impairment (Renal and urinary disorders) | 1 | 1
Ureteric stenosis (Renal and urinary disorders) | 1 | 0
Urethral obstruction (Renal and urinary disorders) | 1 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 7 | 1
Urinary tract disorder (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 4 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Penile swelling (Reproductive system and breast disorders) | 1 | 0
Perineal pain (Reproductive system and breast disorders) | 0 | 1
Scrotal swelling (Reproductive system and breast disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 3
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 | 3
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 42 | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 0
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic aneurysm rupture (Vascular disorders) | 1 | 0
Arterial occlusive disease (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 11 | 3
Hypertension (Vascular disorders) | 7 | 2
Hypertensive crisis (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 4 | 2
Malignant hypertension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 3 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 1
Venous haemorrhage (Vascular disorders) | 1 | 0
Uveitis (Eye disorders) | 1 | 0
Radiculitis (Nervous system disorders) | 0 | 1
Infection (Infections and infestations) | 2 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cabozantinib (N=681) | Prednisone (N=342)
Anaemia (Blood and lymphatic system disorders) | 203 | 111
Thrombocytopenia (Blood and lymphatic system disorders) | 42 | 20
Hypothyroidism (Endocrine disorders) | 94 | 1
Abdominal pain (Gastrointestinal disorders) | 76 | 16
Abdominal pain upper (Gastrointestinal disorders) | 43 | 16
Constipation (Gastrointestinal disorders) | 227 | 100
Diarrhoea (Gastrointestinal disorders) | 349 | 68
Dry mouth (Gastrointestinal disorders) | 65 | 11
Dyspepsia (Gastrointestinal disorders) | 58 | 6
Dysphagia (Gastrointestinal disorders) | 41 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 37 | 7
Nausea (Gastrointestinal disorders) | 390 | 102
Stomatits (Gastrointestinal disorders) | 127 | 8
Vomiting (Gastrointestinal disorders) | 271 | 67
Asthenia (General disorders) | 228 | 63
Fatigue (General disorders) | 338 | 119
General physical health deterioration (General disorders) | 47 | 13
Muscosal inflammation (General disorders) | 134 | 9
Oedema peripheral (General disorders) | 101 | 43
Pain (General disorders) | 56 | 33
Pyrexia (General disorders) | 67 | 36
Urinary tract infection (Infections and infestations) | 71 | 29
Alanine aminotransferase increased (Investigations) | 56 | 10
Aspartate aminotransferase increased (Investigations) | 70 | 14
Weight decreased (Investigations) | 237 | 41
Decreased appetite (Metabolism and nutrition disorders) | 407 | 99
Dehydration (Metabolism and nutrition disorders) | 38 | 15
Hypocalcaemia (Metabolism and nutrition disorders) | 50 | 20
Hypokalaemia (Metabolism and nutrition disorders) | 69 | 9
Hypomagnesaemia (Metabolism and nutrition disorders) | 36 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 91 | 50
Back pain (Musculoskeletal and connective tissue disorders) | 115 | 64
Bone pain (Musculoskeletal and connective tissue disorders) | 109 | 63
Muscle spasms (Musculoskeletal and connective tissue disorders) | 48 | 20
Muscular weakness (Musculoskeletal and connective tissue disorders) | 48 | 22
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 43 | 37
Pain in extremity (Musculoskeletal and connective tissue disorders) | 98 | 36
Dizziness (Nervous system disorders) | 48 | 19
Dysgeusia (Nervous system disorders) | 175 | 16
Headache (Nervous system disorders) | 87 | 14
Depression (Psychiatric disorders) | 42 | 11
Insomnia (Psychiatric disorders) | 53 | 28
Cough (Respiratory, thoracic and mediastinal disorders) | 52 | 15
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 180 | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 135 | 46
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 37 | 9
Dry skin (Skin and subcutaneous tissue disorders) | 53 | 8
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 200 | 5
Hypertension (Vascular disorders) | 191 | 38
Hypotension (Vascular disorders) | 36 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreements with investigators vary; constant is our right to review results communications prior to public release, and embargo communications for a period of ≤60 days from submittal for review. We do not prohibit investigators from publishing, but we may require previously undisclosed confidential information, other than study results, to be removed from publications, and single-center publications are postponed until after publication of the trial's primary multicenter publication.